CLINICAL TRIAL: NCT00008073
Title: Phase I Study Of Octreotide Acetate (Sandostatin) (SMS) As A Biomodulator Of Doxorubicin (DOX)
Brief Title: Octreotide and Doxorubicin in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura A. Pollice, Clinical Research Manager, University of Pittsburgh
Purpose: Treatment
Other Study IDs: 95-088; CDR0000068373 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-951264; NCI-G00-1886
Record Dates: First submitted 2001-01-06; First posted 2004-05-24 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Doxorubicin; Octreotide

INTERVENTIONS:
Drug: doxorubicin hydrochloride
Drug: octreotide acetate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Octreotide may help doxorubicin kill more cancer cells by making tumor cells more sensitive to the drug.

PURPOSE: Phase I trial to study the effectiveness of octreotide and doxorubicin in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and maximum tolerated dose of octreotide administered with doxorubicin in patients with advanced cancer. II. Determine the pharmacokinetics and pharmacodynamics of this treatment regimen in these patients.

OUTLINE: This is a dose escalation study of octreotide. Patients receive doxorubicin IV over 5 minutes on day 1 of course 1. For all subsequent courses, patients receive octreotide SC continuously on days 1-7 and doxorubicin IV over 5 minutes on day 5. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable or responsive disease after 3 courses of therapy receive a maximum of 6 additional courses. Cohorts of 3-6 patients receive escalating doses of octreotide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 21-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignancy ineligible for therapy of proven greater benefit than doxorubicin alone Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL SGOT no greater than 4 times normal Renal: Creatinine no greater than 2 mg/dL Cardiovascular: LVEF at least 50% No compensated or uncompensated congestive heart failure Other: Not pregnant Fertile patients must use effective contraception during and for 2 months after study No history of gallstones with gallbladder in place

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosourea) and recovered No more than 240 mg/m2 total cumulative dose of prior doxorubicin Endocrine therapy: Prior octreotide allowed Recovered from prior octreotide Radiotherapy: At least 3 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-01; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. S. Long, MD, PhD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States